CLINICAL TRIAL: NCT00438789
Title: The Paroxysmal Nocturnal Hemoglobinuria Early Access Treatment Protocol
Acronym: EMBRACE
Status: Approved for marketing | Type: Expanded Access
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Maria Whelden, Alexion Pharmaceuticals
Other Study IDs: C06-002
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2011-09

CONDITIONS: Hemoglobinuria, Paroxysmal
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — eculizumab

INTERVENTIONS:
Drug: eculizumab — 600mg IV every week and 900mg IV every 2 weeks

SUMMARY:
The primary objective is to provide access to eculizumab for PNH patient pending commercial availability.

ELIGIBILITY:
Inclusion Criteria:

* PNH;
* At least 18 years old
* Avoid conception; and
* Willing and able to give written informed consent

Exclusion Criteria:

* Active bacterial infection
* Participation in any other drug trial
* Pregnant breast feeding, or intending to conceive
* Not vaccinated against N meningitidis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Anthony Botti, Livingston, New Jersey, United States